CLINICAL TRIAL: NCT02834832
Title: Novel Coating to Minimize Bacterial Adhesions and Tooth Wear in Denture Acrylic
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600805; UFirst 5154 (Other: UFirst)
Record Dates: First submitted 2016-06-30; First posted 2016-07-15 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Denture Stomatitis; Wear of Denture Teeth
MeSH Terms: conditions — Stomatitis, Denture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: The patients will be given removable dentures with no coatings. These dentures are part of the standard of care to treat their edentulism.
- PECVD Coatings: The patients will be given removable partial dentures with PECVD coatings on both the tissue surface of the dentures and the acrylic denture teeth.
  Interventions: Device: PECVD coating

INTERVENTIONS:
Device: PECVD coating — SiO2/SiC coatings will be applied to the surface of removable partial dentures and denture teeth.
  Groups: PECVD Coatings

SUMMARY:
This study evaluates the effect of coatings on bacterial adhesion on denture acrylic and the wear of denture teeth.

DETAILED DESCRIPTION:
Denture stomatitis is a prevalent disease among removable denture wearers. The cause of this disease stems from a myriad of factors including host immunity and poor oral hygiene. Denture acrylic material is very conducive for the growth and adhesion of bacteria because of its porous nature. The application of plasma enhanced chemical vapor deposited (PECVD) coatings on the surface of acrylic dentures can produce a less porous surface which may minimize the adhesion of bacteria and therefore colonization. The goal is the application of these coatings will help minimize the occurrence of denture stomatitis.

Another issue of removable dentures is the low wear resistance of denture teeth. The application of these coatings on denture teeth should minimize wear of these teeth and prolong the life of removable dentures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are missing some teeth and will need removable dentures

Exclusion Criteria:

* Medical contraindication for dental treatment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seeking care in a Dental Clinic who have removable dentures.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Change in Bacterial Count | 2,4 and 12 weeks
  Biofilms on the tissue surface of the dentures will be obtained for the aforementioned time intervals. Biofilm counts will be analyzed to determine the effect of the coatings on the number of disease causing bacteria on the surface of the denture

SECONDARY OUTCOMES:
wear of denture teeth | 6 months
  Denture teeth will be analyzed for wear at 6 months to determine the effect of PECVD coatings on the wear of denture teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Josephine F. Esquivel-Upshaw, DMD, MS, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No